CLINICAL TRIAL: NCT00987493
Title: Rituximab, Bendamustine and Lenalidomide in Patients With Aggressive B-cell Lymphoma Not Eligible for High Dose Chemotherapy or Anthracycline-Based Therapy. A Phase I/II Trial.
Brief Title: Rituximab, Bendamustine Hydrochloride, and Lenalidomide in Treating Patients With Aggressive B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 38/08; SWS-SAKK-38/08; 2009-012559-67 (EudraCT Number); EU-20976; CDR0000652127
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular | interventions — Rituximab; Bendamustine Hydrochloride; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with rituximab, bendamustine and lenalidomide (Experimental)
  Interventions: Biological: rituximab; Drug: bendamustine hydrochloride; Drug: lenalidomide

INTERVENTIONS:
Biological: rituximab — day 1 at a fixed dose of 375mg/m2
  Other Names: MabThera; Rituxan
Drug: bendamustine hydrochloride — Bendamustine at day 1 and 2 according to the dose escalation in phase I, and at the recommended dose in phase II: 70mg/m2.
  Other Names: Cephalon
Drug: lenalidomide — Lenalidomide at days 1-21 according to the dose escalation in phase I, and at the recommended dose in phase II: 10mg
  Other Names: Revlimid

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer cell growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cell-killing substances to them. Drugs used in chemotherapy, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Lenalidomide may stop the growth of cancer by blocking blood flow to the tumor. Giving rituximab together with bendamustine hydrochloride and lenalidomide may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of giving rituximab together with bendamustine hydrochloride and lenalidomide in treating patients with aggressive B-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum-tolerated dose of the combination of rituximab, bendamustine hydrochloride, and lenalidomide in patients with aggressive B-cell lymphoma not eligible for anthracycline-based first-line treatment or intensive regimens including high-dose therapy (HDT) followed by autologous stem cell transplantation (ASCT) in refractory or relapsing disease, or as treatment for patients relapsing after HDT with ASCT. (phase I).
* To identify the recommended dose of this regimen for a phase II study (phase I).
* To determine the efficacy and safety of this regimen in these patients (phase II).

Secondary

* To assess the quality of life (QOL) of patients treated with this regimen (phase II).
* To evaluate the usefulness and feasibility of the SAKK Cancer-Specific Geriatric Assessment (C-SGA) in patients treated with this regimen (phase II).
* To assess the association between WHO performance status, QOL indicators, and SAKK C-SGA scores (phase II).
* To describe changes in SAKK C-SGA scores from pre- to post-treatment and in QOL (phase II).

OUTLINE: This is a multicenter, phase I dose-escalation study of bendamustine hydrochloride and lenalidomide followed by a phase II study.

Patients receive rituximab IV on day 1, bendamustine hydrochloride IV over 30-60 minutes on days 1-2, and oral lenalidomide on days 1-21. Courses repeat every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients on phase II study complete the SAKK Cancer-Specific Geriatric Assessment at baseline and after completion of course 1. Patients also complete quality-of-life questionnaires at baseline and periodically during study.

After completion of study therapy, patients are followed for up to 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive B-cell non-Hodgkin lymphoma, including any of the following:

  * Diffuse large B-cell lymphoma (variants, subgroups, and subtypes according to WHO criteria)
  * Transformed follicular lymphoma
  * Follicular lymphoma grade 3B
* Meets 1 of the following criteria:

  * Not eligible for anthracycline-based first-line chemotherapy (e.g., R-CHOP)
  * Refractory disease after at least 2 courses of anthracycline-based immune-chemotherapy (e.g., R-CHOP) and patient is not eligible for intensive salvage regimens including HDT with ASCT
  * Relapsed disease after at least 1 treatment with curative intention and patient is not eligible for intensive salvage regimens including HDT with ASCT
  * Relapsed disease after HDT with ASCT
* Measurable disease defined as ≥ 1 lesion ≥ 2 cm in greatest transverse diameter on cross-sectional imaging
* Must complete pre-treatment cancer-specific geriatric assessment and/or quality-of-life questionnaire (phase II only)
* No known CNS involvement

  * Diagnostic procedures required only in case of specific symptoms

PATIENT CHARACTERISTICS:

* WHO performance status (PS) 0-2

  * WHO PS 3 allowed in case of lymphoma-related impaired general condition (phase II only)
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2 times ULN
* Alkaline phosphatase 2 times ULN
* Creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study therapy
* EF ≥ 40% by echocardiography or MUGA scan
* Negative HIV test
* Able to comply with and geographic proximity to allow proper staging and study follow-up
* Agree to follow the special prescribing requirements for lenalidomide
* No other malignancy within the past 3 years except adequately treated cervical carcinoma in situ or localized nonmelanoma skin cancer
* No unstable cardiovascular disease
* No psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent, or interfering with compliance for oral drug intake
* No serious underlying medical condition that, in the judgement of the investigator, could impair the ability of the patient to participate in the trial including, but not limited to, any of the following conditions:

  * Acute or ongoing infection
  * Uncontrolled diabetes mellitus
  * Active autoimmune disease
* No known hypersensitivity to any component of the trial drugs

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No experimental drugs within the past 30 days
* No concurrent drugs contraindicated with the trial drugs according to the Swissmedic-approved product information
* No other concurrent anticancer or investigational drugs or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2009-09; Primary Completion 2014-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (phase I) | at 4 weeks.
Maximum-tolerated dose (phase I) | at the end of phase I (31 August 2011)
Objective response (complete and partial response) (phase II) | phase II (3 years)

SECONDARY OUTCOMES:
Adverse events according to NCI CTCAE v. 3.0 | All AEs will be assessed according to NCI CTCAE v3.0 until 30 days after trial therapy end.
Event-free survival (phase II) | up to 30 months for each patient.
Response duration (phase II) | up to 30 months for each patient.
  From the time when criteria for response (CR/CRu or PR) are met, until documentation of relapse or progression thereafter. Only patients with a response (CR/ CRu or PR) shall be included in this analysis. Patients with no disease progression or relapse shall be censored at the last time they were known to be in remission
Time to progression (phase II) | up to 30 months for each patient.
  Defined as the time from registration until documented lymphoma progression or death as a result of lymphoma. Patients not experiencing an event will be censored at the last time they were known to be in remission
Overall survival (phase II) | up to 30 months for each patient.
Quality of life | approx. 5 months for each patient.
Usefulness and feasibility of the SAKK C-SGA | End of phase II (excluding follow-up) at 3 years.
Association between WHO performance status, QOL indicators, and SAKK C-SGA scores | End of phase II (excluding follow-up) at 3 years.
Progression Free Survival (PFS) | up to 30 months for each patient.
  Time from registration until one of the following events (whichever occurs first):
  * Relapse or progression assessed according to the International Workshop NHL criteria (1999)
  * Death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas Hitz, MD, Principal Investigator — Cantonal Hospital of St. Gallen; Mey Ulrich, MD, Study Chair — Kantonsspital Graubünden
Locations (16):
- Switzerland (16):
  - Kantonsspital Baden, Baden
  - Universitaetsspital Basel, Basel
  - St. Claraspital AG, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Kantonsspital Bruderholz, Bruderholz
  - Kantonsspital Graubünden, Chur
  - Hopital Fribourgeois, Fribourg
  - Hôpitaux Universitaires de Genève HUG, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Stadtspital Triemli, Zurich
  - Universitäts Spital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hitz F, Zucca E, Pabst T, Fischer N, Cairoli A, Samaras P, Caspar CB, Mach N, Krasniqi F, Schmidt A, Rothermundt C, Enoiu M, Eckhardt K, Berardi Vilei S, Rondeau S, Mey U. Rituximab, bendamustine and lenalidomide in patients with aggressive B-cell lymphoma not eligible for anthracycline-based therapy or intensive salvage chemotherapy - SAKK 38/08. Br J Haematol. 2016 Jul;174(2):255-63. doi: 10.1111/bjh.14049. Epub 2016 Mar 28. PMID 27018242
- [Result] Hitz F, Fischer N, Pabst T, Caspar C, Berthod G, Eckhardt K, Berardi Vilei S, Zucca E, Mey U; Swiss Group for Clinical Cancer Research (SAKK), Bern, Switzerland. Rituximab, bendamustine, and lenalidomide in patients with aggressive B cell lymphoma not eligible for high-dose chemotherapy or anthracycline-based therapy: phase I results of the SAKK 38/08 trial. Ann Hematol. 2013 Aug;92(8):1033-40. doi: 10.1007/s00277-013-1751-z. Epub 2013 Apr 17. PMID 23592273